CLINICAL TRIAL: NCT02729129
Title: Face Masks to Reduce the Adverse Effects of Diesel Exhaust Inhalation
Acronym: FM-RADIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: University of Edinburgh (Other)
Responsible Party: Principal Investigator, Jenny Bosson, PhD, MD, Umeå University
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 14-12-31M
Record Dates: First submitted 2016-03-18; First posted 2016-04-06 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: Diesel exhaust; Air pollution; Intervention; Plethysmography

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Commercially available highly-efficient facemask (Experimental)
  Interventions: Other: Diesel exhaust exposure with filtered facemask
- Sham facemask (Sham Comparator)
  Interventions: Other: Diesel exhaust exposure with sham mask

INTERVENTIONS:
Other: Diesel exhaust exposure with filtered facemask — 1 hour exposure to dilute diesel exhaust (approximate particle matter concentration 300 mcg/m3) during intermittent exercise while wearing a filtered facemask.
  Arms: Commercially available highly-efficient facemask
Other: Diesel exhaust exposure with sham mask — 1 hour exposure to dilute diesel exhaust (approximate particle matter concentration 300 mcg/m3) during intermittent exercise while wearing a sham facemask.
  Arms: Sham facemask

SUMMARY:
Air pollution exposure is a major environmental and public health concern. The findings from controlled exposure studies have given biological plausibility to the epidemiological associations, and have defined important pathways that may be amenable to intervention. Ultimately, there is a need to address how one may protect the public from these detrimental effects. Two studies have been performed assessing the cardiovascular effects of wearing a face mask in a highly polluted urban area in China in healthy volunteers and patients with coronary heart disease. These demonstrated lower blood pressure and increased heart rate variability when wearing a face mask as compared to not. The investigators aim to test if wearing a highly efficient face mask during exposure to dilute diesel exhaust abrogates the well-known adverse cardiovascular effects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Non-smoking
* All subjects undergo a general health examination and are required to have normal clinical examination, ECG, blood tests and lung function

Exclusion Criteria:

* Metabolic or cardiovascular disease
* Asthma or other respiratory disease
* Respiratory infection within 2 weeks of the study
* Antioxidant- and/or vitamin supplementation within 1 week prior to, as well as during the course of the study. (incl vitamin C, Acetylcysteine)
* Smokers or regular snus usage

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2014-04; Primary Completion 2015-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Vascular vasomotor function | 2 hours
  Forearm venous occlusion plethysmography to measure forearm blood flow during unilateral intrabrachial infusion of endothelial-dependent and -independent vasodilators. Assessment is shown in ml/100ml tissue/min.

SECONDARY OUTCOMES:
Fibrinolytic function | 2 hours
  Tissue plasminogen activator was analysed in blood samples taken after bradykinin infusions in order to assess fibrinolytic function (ng/ml).
Blood pressure | 24 hours
  Ambulatory blood pressure monitors are worn by subjects for 24 hours during and after exposure.
Heart rate variability | 24 hours
  Holter ECGs are worn by subjects during and for 24 hours post exposure. This will be assessed for heart rate variability (HRV).

CONTACTS AND LOCATIONS:
Overall Officials: Jenny A Bosson, MD, PhD, Principal Investigator — Umeå University
Locations (1):
- Umeå University, Umeå, Sweden